CLINICAL TRIAL: NCT00816686
Title: A Phase 1, Open-Label, Multi-center, Dose Escalation Study of the Safety and Pharmacokinetics of AGS-16M18 Given as Monotherapy in Subjects With Advanced Renal Cell Carcinoma
Brief Title: A Phase 1 Study of the Safety and Pharmacokinetics of AGS-16M18 in Subjects With Advanced Renal Cell Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial was terminated due to the need to re-formulate the study drug.
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007002
Record Dates: First submitted 2009-01-01; First posted 2009-01-05 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2010-05

CONDITIONS: Carcinoma, Renal Cell; Kidney Neoplasms; Kidney Diseases
Keywords: clinical trial, phase 1; carcinoma, advanced renal cell; kidney; pharmacokinetics; safety; AGS-16M18
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Kidney Diseases; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1. AGS-16M18 Dose 1 (Experimental)
  Interventions: Biological: AGS-16M18
- 2. AGS-16M18 Dose 2 (Experimental)
  Interventions: Biological: AGS-16M18
- 3. AGS-16M18 Dose 3 (Experimental)
  Interventions: Biological: AGS-16M18
- 4. AGS-16M18 Dose 4 (Experimental)
  Interventions: Biological: AGS-16M18
- 5. AGS-16M18 Dose 5 (Experimental)
  Interventions: Biological: AGS-16M18

INTERVENTIONS:
Biological: AGS-16M18 — IV Infusion

SUMMARY:
This is a first in human study of AGS-16M18 given every week to subjects with advanced renal cell cancer. AGS-16M18 will be administered as a 60 minute IV infusion on consecutive days until the disease worsens.

DETAILED DESCRIPTION:
Subjects will be enrolled sequentially into 5 planned dose cohorts according to a standard, dose escalation study design. A disease assessment will be performed at study week 5 (+/- 3 days) by the investigator. The assessment will be based both on changes in clinical symptoms, and radiographic images. Subjects without evidence of disease progression may receive AGS-16M18 extended therapy at the dose and schedule of their assigned cohort until disease progression or intolerability of AGS-16M18. Disease assessments will be performed every 8 weeks during the extended period. A safety follow-up visit will occur 4 weeks after the last infusion of AGS-16M18.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis (recent or remote) of metastatic renal cell carcinoma (including papillary, clear cell, and excluding transitional cell types) that is not amendable to cure by surgery or other means, and must have failed at least one prior systemic therapy, including but not limited to treatment with sunitinib, temsirolimus or sorafenib
* Evaluable/Measureable disease according to Response Criteria for Solid tumors
* Eastern Cooperative Group performance status of 0-1
* Therapeutic anti-coagulation (PT, and/or INR, PTT) permitted, if clinically stable and >/= 3 months from initiation

Exclusion Criteria:

* Past or present documented central nervous system (CNS) tumor or CNS metastasis
* Use of investigational drug (including marketed drugs not approved for this indication) within 4 weeks prior to screening or 5 half-lives of the prior investigational drug (whichever is longer)
* History of thromboembolic events and bleeding disorders </= 3 months (e.g., DVT or PE)
* Major Surgery (that requires general anesthesia) within 4 weeks of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Throughout the treatment
Assessment of PK variables | Weeks 0 - 5, week 8, weekly during extension period, 2 and 3 months after last dose

SECONDARY OUTCOMES:
Incidence of anti-AGS-16M18 antibody formation | Week 0, week 1, week 4, week 8, every 8 weeks during extension period, 2 and 3 months after last dose
Changes in tumor status | Week 5, week 8, every 8 weeks during extension period

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Agensys, Inc.
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - New York, New York